CLINICAL TRIAL: NCT01639859
Title: Assessment of Supersonic Imagine Aixplorer for the Detection and Localisation of Prostate Cancer Foci
Acronym: PROSTATE SSI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2011.658
Record Dates: First submitted 2012-06-22; First posted 2012-07-13 (Estimated); Last update posted 2025-01-10 (Actual); Status verified 2025-01

CONDITIONS: Cancer of Prostate
Keywords: prostate cancer; elastography; elasticity
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Elastography (Experimental)
  Interventions: Other: Elastography

INTERVENTIONS:
Other: Elastography — The elastography in vivo will be performed before the prostatectomy. The elastography ex vivo will be performed after radical prostatectomy.
  Other Names: Supersonic Imagine Aixplorer scanner

SUMMARY:
The primary aim of the study is to assess the elasticity (Young's modulus) of cancerous tumor foci, of normal peripheral zone, and of normal transition zone in the prostate. Images obtained with the Supersonic Imagine Aixplorer scanner prior to radical prostatectomy are compared to whole-mount histology.

ELIGIBILITY:
Inclusion Criteria:

* Patient over 18 years old, with prostate cancer and scheduled for radical prostatectomy

Exclusion Criteria:

* Medical history of prostate surgery or radiotherapy of prostate
* Medical history of abdominal perinéanal amputation or whole of state which prevent to use endorectal probe

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2011-10; Primary Completion 2012-10 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Young's modulus(kPa) of cancerous tumor foci | 2 years
Young's modulus(kPa) of normal peripheral zone | 2 years
Young's modulus(kPa) of normal transition zone | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: ROUVIERE Olivier, Pr, Principal Investigator — Hospices Civils de Lyon
Locations (1):
- Service de Radiologie, Pavillon P Radio, Hôpital Edouard Herriot, Lyon, LYON, France

REFERENCES:
- [Background] Rouviere O, Melodelima C, Hoang Dinh A, Bratan F, Pagnoux G, Sanzalone T, Crouzet S, Colombel M, Mege-Lechevallier F, Souchon R. Stiffness of benign and malignant prostate tissue measured by shear-wave elastography: a preliminary study. Eur Radiol. 2017 May;27(5):1858-1866. doi: 10.1007/s00330-016-4534-9. Epub 2016 Aug 23. PMID 27553936